CLINICAL TRIAL: NCT05618106
Title: Modification of the Low FODMAP Diet in Treatment of Irritable Bowel Syndrome: A Randomised Cross-over Study
Brief Title: Low FODMAP Diet in Patients With IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jens Rikardt Andersen (Other)
Responsible Party: Sponsor-Investigator, Jens Rikardt Andersen, Assoc Prof, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FODMAP
Record Dates: First submitted 2022-11-08; First posted 2022-11-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: Carbohydrates; low FODMAP diet; components in the low FODMAP diet
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — FODMAP Diet

STUDY DESIGN:
Intervention Model Description: Cross-over of 3 variations of the low FODMAP diet excluding 1 of the 3 components in every period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- low FODMAP diet (Experimental): Diet low in all kinds of FODMAPS
  Interventions: Other: Low FODMAP DIET = Diet with Low polyol, FOS and GOS
- Low Fodmap diet but polyols allowed (Placebo Comparator): Diet low in FOS and GOS
  Interventions: Other: Low FODMAP DIET = Diet with Low polyol, FOS and GOS
- Low Fodmap diet but FOS and GOS allowed (Active Comparator): Diet low in polyols
  Interventions: Other: Low FODMAP DIET = Diet with Low polyol, FOS and GOS

INTERVENTIONS:
Other: Low FODMAP DIET = Diet with Low polyol, FOS and GOS — Low Polyol diet

SUMMARY:
The aim was aimed to investigate if all carbohydrate groups eliminated in the Low FODMAP diet are equally important in relieving gastrointestinal symptoms in IBS.

in a randomized cross-over design to three different carbohydrate-modified diets: A) Low Polyol diet, B) Low FOS+GOS diet, and C) Low FODMAP diet for three months without wash-out-periods. Gastrointestinal symptoms, Quality of life was measured at baseline and after each intervention diet.

DETAILED DESCRIPTION:
Low FODMAP diets contain 3 major types of carbohydrates to be avoided. The clasical diet is very difficult to maintain over longer periods of time. Therefore, we aimed to investigate if all carbohydrate groups in the Low FODMAP diet are equally important in relieving gastrointestinal symptoms in IBS.

Patients diagnosed with IBS according to the Rome III criteria were randomised in a cross-over design to three different carbohydrate-modified diets: A) Low Polyol diet, B) Low FOS+GOS diet, and C) Low FODMAP diet for a total of three months without wash-out-periods. Gastrointestinal symptoms were assessed by the Birmingham IBS questionnaire and adequate relief (IBS-AR). Quality of life was measured by the IBS Quality of Life Scale questionnaire (IBS-QOL). All registrations were performed at baseline and after each intervention diet.

ELIGIBILITY:
Inclusion Criteria:

* IBS diagnosed by the Rome III criteria and
* referred to the clinic for treatment by diet

Exclusion Criteria:

* Dementia
* lack of ability to speak Danish
* additional chronic diseases prevailing participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Birmingham IBS questionnaire and adequate relief (IBS-AR). | 3 months
  Score in points (low score means few symptoms)

SECONDARY OUTCOMES:
IBS Quality of Life Scale questionnaire (IBS-QOL) | 3 months
  Score in points (high score means better life satisfaction)

CONTACTS AND LOCATIONS:
Overall Officials: Jens R Andersen, MD, MPA, Study Chair — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jensen LG, Kjaer M, Andersen JR. Modification of the Low FODMAP Diet Is Feasible in the Treatment of Irritable Bowel Syndrome: A Randomised Crossover Study. Gastroenterol Res Pract. 2025 Nov 13;2025:4152978. doi: 10.1155/grp/4152978. eCollection 2025. PMID 41278484